CLINICAL TRIAL: NCT04739241
Title: Is Premixed Insulin Therapy an Alternative to Basal Bolus Therapy in Type 2 Diabetes Mellitus People Older Than 65 Years Old: A Pilot Randomised Trial
Brief Title: Premixed vs Basal Bolus Insulin Therapy in Older Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/11
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: premixed insulin therapy; basal-bolus insulin therapy; type 2 diabetes; elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (experimental arm) (Experimental): Premixed insulin therapy
  Interventions: Drug: premixed insulin therapy
- Group B (active comparator) (Active Comparator): Basal bolus insulin therapy
  Interventions: Drug: basal bolus insulin therapy

INTERVENTIONS:
Drug: premixed insulin therapy — Premixed insulin treatment: 30% of the calculated dose was administered before breakfast and before lunch (biphasic insulin lispro 50% or biphasic insulin aspart 50%) and the remaining 40% of the dose before dinner (biphasic insulin lispro 25% or biphasic insulin aspart insulin 30%).
  Arms: Group A (experimental arm)
Drug: basal bolus insulin therapy — Basal-bolus insulin treatment: 50% dose in insulin glargine and 50% dose in insulin lispro or aspartic, distributed in equal parts in the 3 main meals
  Arms: Group B (active comparator)

SUMMARY:
The purpose of this study is to compare efficacy and security of premixed insulin treatment vs basal bolus insulin treatment in older patients with poorly controlled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Age ≥ 65 years old
* Type 2 diabetes mellitus
* HbA1c ≥9% (74 mmol/mol)
* Previously treated with one or two doses of basal insulin and oral hypoglycaemic agents

Exclusion Criteria:

* Severe insulin-resistance
* High doses of corticosteroids
* Chemotherapy treatment
* High comorbidity
* Bad compliance of the treatment
* Frequent severe hypoglycaemia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels | 12 months after recruitment
  Change from baseline in HbA1c levels after 12 months of therapy

SECONDARY OUTCOMES:
Incidence of hypoglycaemia as an adverse effect of the treatment | every month during the 12-month follow-up
  Number of hypoglycaemias by month
Incidence of dosing errors as a measure of the safety of the treatment | every month during the 12-month follow-up
  Number of dosing errors by month
Change in the scores of the Diabetes Treatment Satisfaction Questionnaire (DTSQ) from recruitment to month 12. | 12-month follow-up
  Change from baseline to12 months of therapy using the DTSQ questionnaire of satisfactions with the treatment of diabetes.
Change in the scores of the Diabetes Quality Of Life Questionnaire (EsDQOL) from recruitment to month 12. | 12-month follow-up
  Change from baseline to12 months of therapy using the EsDQOL questionnaire of quality of life in diabetic patients

IPD SHARING:
Plan to Share IPD: No